CLINICAL TRIAL: NCT05063721
Title: Assess Safety of Intra-arterial Autologous Myogenic Stem Cell Therapy for m.3243A>G Mutation Carriers
Brief Title: MABs Therapy m.3243A>G Mutation Carriers
Acronym: MABS01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL68732.000.19
Record Dates: First submitted 2021-07-19; First posted 2021-10-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Mitochondrial Myopathies
Keywords: m.3243A>G; mesoangioblasts
MeSH Terms: conditions — Mitochondrial Myopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-arterial delivery of autologous MABs (Experimental): Autologous mesoangioblasts (MABs) will be intra-arterially delivered to lower leg of participant
  Interventions: Biological: autologous mesoangioblasts
- No intervention (No Intervention): intra-subject control

INTERVENTIONS:
Biological: autologous mesoangioblasts — intra-arterial administration of autologous mesoangioblasts in lower leg (50x10E6/kg)
  Arms: Intra-arterial delivery of autologous MABs

SUMMARY:
Rationale: Mitochondrial disorders are progressive, often fatal multisystem disorders, in 20-25% of the cases caused by heteroplasmic mutations in the mitochondrial DNA (mtDNA). At this moment, there is no effective treatment known to influence the disease process or manifestation. Myogenic stem cell-based therapies complementing defective muscle cells and fibres, are highly promising to combat the myopathy and exercise intolerance which affect >50% of heteroplasmic mtDNA mutation carriers. Myogenic stem cells called mesoangioblasts (MABs), are currently the only myogenic precursors that fulfil all criteria to be used as advanced therapy medicinal product (ATMP) for systemic treatment. The researchers have demonstrated that MABs of most m.3243A>G carriers contain no or only a low amount (<10%) of the mtDNA mutation, allowing direct ex vivo expansion of patient-derived MABs. The overall aim is to induce muscle regeneration using these autologous MABs with a mutation load of <10%, as an advanced therapy medicinal product (ATMP).

Objective: The phase I trial will consist of an intra-arterial injection (via catheter in femoral artery) of the autologous MABs in the left lower leg of 5 m.3243A>G patients.

DETAILED DESCRIPTION:
Rationale: Mitochondrial disorders are progressive, often fatal multisystem disorders, in 20-25% of the cases caused by heteroplasmic mutations in the mitochondrial DNA (mtDNA). Epidemiological studies have shown that mtDNA disorders affect about 1 in 10,000 of the general population, inducing significant morbidity and mortality and high health and societal costs. Clinical manifestations are most prominent in organs with a high energy demand, like muscle and brain. At this moment, there is no effective treatment known to influence the disease process or manifestation. Myogenic stem cell-based therapies complementing defective muscle cells and fibres, are highly promising to combat the myopathy and exercise intolerance which affect >50% of heteroplasmic mtDNA mutation carriers. Myogenic stem cells called mesoangioblasts (MABs), are currently the only myogenic precursors that fulfil all criteria to be used as advanced therapy medicinal product (ATMP) for systemic treatment, namely good ex vivo proliferation capacity, high myogenic capacity and a capability to cross blood vessels, allowing intra-arterial (systemic) delivery towards affected muscle. Both genetically corrected autologous and allogeneic MABs transplantation has been performed in mice and dog models, but only allogeneic MABs transplantation has been performed in patients with Duchene muscular dystrophy (DMD). Treatment with ex-vivo expanded MABs resulted in significant regeneration of DMD positive muscle fibers in both mice and dog models. Intra-arterial delivery of allogeneic MABs in DMD boys (phase I/IIa clinical study) demonstrated that the treatment was relatively safe, and that some dystrophin was produced by the new muscle fibers, although not sufficient for functional improvement. The approach of this study has key advantages as autologous MABs are used, which do not require an immunosuppressive regime. Also, mitochondrial function is partly preserved in mtDNA mutation carriers and partial supplementation by healthy fibres should suffice to ameliorate mitochondrial function. The researchers have demonstrated that MABs of most m.3243A>G carriers contain no or only a low amount (<10%) of the mtDNA mutation, allowing direct ex vivo expansion of patient-derived MABs. The overall aim is to induce muscle regeneration using these autologous MABs with a mutation load of <10%, as an advanced therapy medicinal product (ATMP). This proposal covers the first phase I/IIa trial.

Objective: The phase I/IIa trial will consist of an intra-arterial injection (via catheter in femoral artery) of the autologous MABs in the left lower leg of 5 m.3243A>G patients. The primary objective is assessing safety of administration of autologous MABs, which have not been used as treatment before in humans. Secondary objectives are (1) to assess homing of the labelled autologous MABs to the tibialis anterior muscle 24 hours after i.a. delivery, and (2) assess effectiveness at the tissue level by measuring myogenesis and mtDNA mutation load of treated tibialis anterior muscle compared with untreated muscle from the contralateral leg.

Study design: Mono-center prospective open label intra-subject controlled phase I/IIa clinical study.

Study population: 15 adult m.3243A>G patients, of which 5 will be enrolled in the clinical study.

Intervention: All 15 adult m.3243A>G patients will undergo a ~30mg m. vastus lateralis muscle biopsy at visit 1. From these 15 patients, five patients will enroll the clinical study based on their m.3243A>G mutation load in skeletal muscle and mesoangioblasts. These 5 patients will visit the MUMC for four additional times. From each patient, during visit 2 till 5, in total five muscle biopsies will be collected (1x ~100 mg m.vastus lateralis both legs at visit 2, 2x ~30mg m. tibialis anterior both legs at visit 4 and 2x ~30mg m. tibialis anterior both legs at visit 5). At visit 4, the tibialis anterior muscle of one leg will be treated with 5*10E7/kg autologous MABs via tibial anterior artery delivery. A bout of maximal eccentric exercise will be executed at visit 3. Venous blood samples will be taken at all visits.

Main study parameters/endpoints: The primary endpoint is to assess safety will be by monitoring infusion (angiography), monitoring for acute adverse effects (24hrs), blood sampling and muscle sampling to assess local and systemic inflammation and muscle markers (CK). Secondary endpoints are assessment of effectiveness at the tissue level: namely, migration of the IC-Green labelled mesoangioblasts from the bloodstream into the tibialis anterior muscle (24 hrs after infusion) and formation of new muscle fibers and m.3243A>G mutation load (28 days after infusion).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Out of the 15 patients, 5 patients will enrol the clinical study and visit the hospital five times in total. The 10 patients, who are not selected, will visit the MUMC once.

* At the first visit (all 15 patients), a neurological and routine clinical examination and one vastus lateralis skeletal muscle biopsy (~30mg) will be collected.
* At the second visit (5 patients), a routine physical examination will be performed, and a vastus lateralis skeletal muscle biopsy (~100mg) and a venous blood sample (~10 ml) will be collected and they will try-out the bout of eccentric exercise.
* At visit 3: routine physical examination, a bout of maximal eccentric exercise will be performed and a venous blood sample (10ml) will be collected.
* At visit 4: routine physical examination, intra-arterial administration of 5*10E7 MABs in one leg, followed by 24hrs observation in the hospital including regular blood sampling (4x ~10ml) and a ~30mg tibialis anterior muscle biopsy of both legs 24 hours after infusion of the autologous MABs.
* Visit 5 consists of a neurological and routine physical examination, a venous blood sample (~10ml) and a ~30mg muscle biopsy in the tibialis anterior muscles of both legs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age: 18+
* Sex: male/female
* Patients with the m.3243A>G mutation

Exclusion Criteria:

* Use of anti-coagulants, anti-thrombotics and other medication influencing coagulation
* Have a weekly alcohol intake of ≥ 35 units (men) or ≥ 24 units (women)
* Current history of drug abuse
* Deficient immune system or autoimmune disease
* Significant concurrent illness
* Ongoing participation in other clinical trials
* Major surgery within 4 weeks of the visit
* Vaccination within 4 weeks of the visit
* Pregnant or lactating women
* Psychiatric or other disorders likely to impact on informed consent
* Patients unable and/or unwilling to comply with treatment and study instructions
* Any other factor that in the opinion of the investigator excludes the patient from the study
* A history of strokes
* Allergy for contrast fluid
* Peripheral signs of ischemia or vasculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Assess blood flow in lower leg following intra-arterial delivery of autologous MABs as ATMP. | Day 1, directly after ATMP administration
  Assess blood flow in lower leg using digital subtraction angiography (DSA).
Assess adverse events following intra-arterial delivery of autologous MABs as ATMP in one lower leg. | 1 month
  Assessment of adverse events
Assess systemic inflammation following intra-arterial delivery of autologous MABs as ATMP in one lower leg. | Day 1
  Analysis inflammation markers blood (IL6, TNFa, CK)
Assess systemic inflammation following intra-arterial delivery of autologous MABs as ATMP in one lower leg. | Day 28
  Analysis inflammation markers blood (IL6, TNFa, CK)
Assess local inflammation following intra-arterial delivery of autologous MABs as ATMP in one lower leg. | Day 1
  Analysis inflammation markers (IL6, TNFa, CK) in tibialis anterior muscle
Assess local inflammation following intra-arterial delivery of autologous MABs as ATMP in one lower leg. | Day 28
  Analysis inflammation markers (IL6, TNFa, CK) in tibialis anterior muscle

SECONDARY OUTCOMES:
Assess preliminary effectiveness based on MABs homing to the tibialis anterior muscle | Day 1
  Determine the number of IC-Green positive MABs per mg muscle tissue by measuring the near infrared signal on a Licor Odessey CLx of the tibialis anterior muscle biopsies of the infused and not-infused leg, and a dilution series of IC-Green labeled MABs.
Assess preliminary effectiveness based on MABs-induced myogenesis | Day 28
  Determine the numbers of NCAM+ muscle fibers per field in the muscle biopsy of the treated tibialis anterior muscle compared with the muscle biopsy of the non-injected contra lateral tibialis anterior muscle.
Assess preliminary effectiveness based on changes in mtDNA mutation load in newly formed muscle fibers | Day 28
  Determine the m.3243A>G mutation load by Genescan fragment analysis of laser capture micro-dissected NCAM+ fibers from the tibialis anterior muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Faber, Prof. PhD MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Tienen F, Zelissen R, Timmer E, van Gisbergen M, Lindsey P, Quattrocelli M, Sampaolesi M, Mulder-den Hartog E, de Coo I, Smeets H. Healthy, mtDNA-mutation free mesoangioblasts from mtDNA patients qualify for autologous therapy. Stem Cell Res Ther. 2019 Dec 21;10(1):405. doi: 10.1186/s13287-019-1510-8. PMID 31864395